CLINICAL TRIAL: NCT00908843
Title: Comparative Efficacy of the Application of an Oral/iv Hydration Protocol in the Prevention of Contrast Induced Nephropathy
Brief Title: Prevention of Contrast Induced Nephropathy (NIC) by Intravenous Versus Oral Rehydration
Acronym: NIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIC2117; 2117/2007; EC08/00203
Record Dates: First submitted 2009-05-25; First posted 2009-05-27 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: KIDNEY FAILURE, ACUTE
Keywords: Contrast nephropathy; Renal failure
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency | interventions — Bicarbonates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- (I) BICARBONATE INTRAVENOUS INFUSION (Experimental): Intravenous hydration with bicarbonate 1/6 M intravenous infusion (3ml/Kg/h) one hour before the administration of intravenous contrast
  Interventions: Other: Intravenous hydration with bicarbonate
- (II) ORAL SODIUM SOLUTION (Active Comparator): Oral hydration with Sodium solution (Casen solution of rehydratation) in the 4 hours before of the intravenous contrast administration (75 ml/10 kg as equivalent to 0,25 g of sodium chloride /10 kg).
  Interventions: Other: Oral hydration with Sodium solution

INTERVENTIONS:
Other: Intravenous hydration with bicarbonate — Intravenous hydration with bicarbonate 1/6 M intravenous infusion (3ml/Kg/h) one hour before the administration of intravenous contrast
  Arms: (I) BICARBONATE INTRAVENOUS INFUSION
Other: Oral hydration with Sodium solution — Oral hydration with Sodium solution (Casen solution of rehydration) in the 4 hours before of the intravenous contrast administration (75 ml/10 kg as equivalent to 0,25 g of sodium chloride /10 kg).
  Arms: (II) ORAL SODIUM SOLUTION

SUMMARY:
The purpose of this study is to compare the efficacy of oral versus intravenous hydration in the prevention of the contrast-induced nephropathy.

DETAILED DESCRIPTION:
Objective: To compare the efficacy of oral versus intravenous hydration in the prevention of the contrast-induced nephropathy (CIN) in inpatients with different renal function and equal type and volume of contrast.

Methods: The clinical trial will include 324 patients with GFR higher or equal to 30 ml/min who will receive intravenous contrast (Iohexol: 300 mg of l/ml; approximate volume: 120 ml at 2-5ml/second) in the following 12-24 hours. Patients with inclusion criteria, and having previously signed a consent form, will be randomised into 3 groups (intravenous hydration, oral and no hydration). Intravenous hydration will be carried out with bicarbonate 1/6M one hour before the test (3ml/Kg/h) and oral hydration with Casen solution in will be carried out 4 hours before (75 ml/10 kg) the intravenous contrast administration. In relation to the hydrated, it should be pointed out that, the same procedure would have been carried out without the study. The follow-up of renal function will be carried out after measuring creatinine and cystatin C in blood and GFR pre- and 24 hour after the test. It will also determine neutrophil gelatinase-associated lipocalin (N-GAL), IL-8 and F2-Isoprostanes levels in urine and superoxide dismutase activity in erythrocytes, pre- and in different post- test times.

Also, in vitro, the effect of contrast on NADPH-oxidase activity of PBLs isolated from 30 control patients will also be studied (10 patients by each group).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients
* aged less than 18 years
* provision for the performance of IV contrast (120-150 ml) within 12-24 h.

Exclusion Criteria:

* Nephropathy patients with stage 4-5 according to the classification of Chronic Kidney Disease (CKD) of the U.S. National Kidney Foundation's Kidney Disease Outcome Quality Initiative (NKF-KDOQI). The GFR is estimated by the formula Modification Diet Renal Diseases Study (MDRD).
* Patients undergoing: cardiac catheterization or other proceeding in contrast with the previous week, colonoscopy in 48 hours or have received prior nephrotoxic (aminoglycosides and / or certain chemotherapeutic agents) 24-48 hours before the test or in hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of oral versus intravenous hydration in the prevention of the contrast-induced nephropathy (CIN) in inpatients with different renal function. | 24 h

SECONDARY OUTCOMES:
Study in vitro, the effect of contrast on NADPH-oxidase activity of PBLs isolated from 30 patients will be included in the study (10 patients by each group). | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Nuria García-Fernández, MD, Ph.D., Study Director — Clínica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain